CLINICAL TRIAL: NCT00808041
Title: Breast Cancer Chemotherapy Monitoring With Dedicated Breast Computed Tomography
Brief Title: Chemotherapy Monitoring With Breast Computed Tomography (CT)
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Ioannis Sechopoulos, Ph.D., Assistant Professor of Radiology and Imaging Sciences, Emory University
Other Study IDs: IRB00012068; 1P50CA128301-01A1 (NIH)
Record Dates: First submitted 2008-12-12; First posted 2008-12-15 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: Breast Cancer
Keywords: Neoadjuvant Treatment; Therapy Response; Breast Computed Tomography
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Treatment: Breast cancer patients undergoing hormonal therapy before surgery.
  Interventions: Device: Dedicated breast computed tomography imaging

INTERVENTIONS:
Device: Dedicated breast computed tomography imaging — Pre- and post-contrast enhancement acquisition of breast CT images of tumor-containing breast every two months.
  Other Names: Koning CBCT,Cone Beam Breast CT

SUMMARY:
The purpose of this study is to determine if dedicated breast computed tomography can be used successfully to monitor tumor response in breast cancer patients undergoing neoadjuvant chemotherapy.

DETAILED DESCRIPTION:
Before undergoing surgery to remove the tumor, it is common for breast cancer patients to first undergo chemotherapy or hormonal therapy. The main goal of the therapy is to reduce the size of the tumor before it is removed. Unfortunately, therapy response varies a lot between patients. The development of an effective therapy response monitoring method could reduce the time that a patient undergoes ineffectual therapy or unnecessary therapy after complete response.

Dedicated breast computed tomography (or breast CT), a new way of imaging the breast, has been introduced in the last few years. Breast CT is an x-ray exam that uses 3D imaging to show the breast in its real three dimensional shape. Combined with the use of special chemicals called iodine contrast enhancement, breast CT can provide images of both the anatomy and the blood flow in the breast. We propose to use breast CT to carefully monitor the response to therapy of breast cancer patients undergoing therapy before surgery.

ELIGIBILITY:
3.1 Eligibility Criteria

* All subjects will be women at least 18 years of age that will undergo standard or research pre-operative hormonal therapy for breast cancer before lumpectomy or mastectomy.
* Women who have undergone pre treatment breast MR imaging to verify that no additional findings are present.

3.2 Ineligibility Criteria

* Subject does not meet any of the inclusion criteria
* Women with suspected or confirmed pregnancy
* Women who have had bilateral mastectomy
* Women who are unable to remain in a prone position on the BCT system for the required amount of time
* Women who cannot give informed consent
* Women with metastasis
* Male subjects
* Women with implants
* Women with breast augmentation, except for unilateral augmentation done for prior mastectomy
* Women who are allergic to iodine
* Women with physical limitations such as, but not limited to: frozen shoulder, recent heart surgery, pace maker, neck problems or any other condition that would prohibit them from lying face down
* Women who have had problems or reactions to contrast, such as nausea/vomiting, itching, hives, B/P changes, respirator distress, cardiac arrest.
* Women with history of Diabetes, kidney disease, kidney surgery, dialysis, heart disease-such as Congestive Heart Failure, Multiple Myeloma, Sickle Cell Anemia, Lupus, Rheumatoid Arthritis or other Autoimmune disease, recent surgery, chemotherapy, dehydration, high use of NSAIDs such as Ibuprofen

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population for this study is women who will undergo pre-operative hormonal therapy for breast cancer before lumpectomy or mastectomy.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2009-07; Primary Completion 2012-09 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Tumor response | Mid-treatment and post-treatment completion

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis Sechopoulos, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University Winship Cancer Institute, Atlanta, Georgia, United States